CLINICAL TRIAL: NCT07319312
Title: Evaluating the Clinical Effectiveness and Implementation Outcomes of Nurse-Led Stroke Transitional Care Model in Tanzania
Brief Title: Evaluating the Effect of Nurse-Led Stroke Transitional Care in Tanzania
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Nyagwaswa Athanas Michael, Principal Investigator, Shandong University
Other Study IDs: Shandong@2025; 72274110 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-11-19; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Stroke Acute; Stroke (CVA) or Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Historical control group: Stroke survivors and their caregivers received usual care
  Interventions: Behavioral: Nurse-led stroke transitional care program

INTERVENTIONS:
Behavioral: Nurse-led stroke transitional care program — Participants in intervention group will receive usual care plus nurse-led stroke transitional care. Two nurse champions will conduct the face-to-face sessions while other two nurse researchers will conduct the telephone call sessions between August and December, 2025. During hospitalization, the two nurse champions will conduct five face-to-face sessions (2 individual sessions at admission; and at discharge), and three group sessions with 2-4 dyads of patients and caregivers. After hospitalization, two nurse researchers will conduct seven follow-up sessions for three months via phone calls at day 3, week 1, week 3, week 5, week 7, week 9, and week 11. The face-to-face sessions and phone call sessions will take 40-60 minutes and 20-30 minutes respectively

SUMMARY:
The goal of this observational study is to assess the effects of nurse-led stroke transitional care in stroke survivors, caregivers and healthcare providers who participate in nurse-led stroke transitional care program to improve discharge preparedness, disease self-management and quality of life among stroke survivors. The main question it aims to answer is: does nurse-led stroke transitional care program improve discharge preparedness, disease self-management and quality of life among stroke survivors? Participants are currently participating in nurse-led stroke transitional care program as part of their medical care. Stroke survivors and their caregivers will be followed for six months period to assess their transitional care quality and clinical outcome measures.

ELIGIBILITY:
Inclusion criteria

* Clinical nurses and physicians with six months of working experience in stroke care
* Clinical nurses and physicians with a minimum of diploma in their professions.
* Stroke survivors with 18 years old and above
* Stroke survivors admitted in the stroke units
* Stroke survivors with primary diagnosis of stroke confirmed by brain CT/MRI
* Stroke survivors who undergo usual discharge process
* Stroke survivors who live with their family caregivers
* Stroke survivors who have mobile phones
* Stroke survivors who can read and write
* Stroke survivors who are able to communicate
* Stroke survivors with National Institutes of Health Stroke Scale (NIHSS) < 6
* Stroke survivors with Modified Barthel Index (MBI) > 9
* Stroke survivors with Modified Rankin Scale (mRS) < 5
* Stroke survivors with Montreal Cognitive Assessment Test (MoCA) > 14
* Stroke survivors who are expected to stay in the ward for 3-5 days,
* Stroke survivors who are expected to survive for 3 months
* Family caregivers with mobile phones
* Family caregivers who can read and write
* Family caregivers who are able to communicate
* Family caregivers who live with the patient after stroke

Exclusion criteria

* Healthcare providers who will be on leave during the study period.
* Stroke survivors with previous stroke who are not admitted in stroke units
* Stroke survivors who are discharged against medical advice
* Stroke survivors who have end-stage organ failure
* Stroke survivors who have family caregivers
* Stroke survivors who can't read/write
* Stroke survivors who have no mobile phones.
* Family caregivers without mobile phone that is accessible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include nurses, doctors, stroke survivors and caregivers who are directly involved in hospital-to-home transition.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy among stroke survivors | 6 months after discharge
  Ability to take control and perform recommended health behaviors and discharge instructions. Self-efficacy will be measured by the Stroke Self-Efficacy Questionnaire (a=0.9) developed by Jones and colleagues. This will be measured by a scale as total scores and mean scores. High total and mean scores indicate better ability to follow and adhere to healthy lifestyles after stroke
Quality of life among stroke survivors | 6 months after discharge
  Quality of life that will be measured by the Stroke Specific Quality of Life (SSQoL) with (a=0.85). This will be measured by a scale as total scores and mean scores. High total and mean scores indicate better quality of life as evidenced by ability to perform self-care activities, improved cognitive function, mobility, and engaging in social activities
Discharge preparedness among survivors | within 1 month after discharge
  Discharge preparedness that will be measured by the Short Forms of the Readiness for Hospital Discharge Scale (RHDS) developed by Weiss. This will be measured by a scale as total scores and mean scores. High total and mean scores indicate readiness for hospital-to-home discharge among stroke survivors.
Discharge preparedness among health care providers | within 1 month after discharge
  Discharge preparedness that will be measured by the Short Forms of the Readiness for Hospital Discharge Scale (RHDS) developed by Weiss. This will be measured by a scale as total scores and mean scores. High total and mean scores indicate agreement on readiness for hospital-to-home discharge among nurses and doctors.
Resilience among caregivers | 6 months after discharge
  Resilience will be measured by the 10-items Connor-Davidson Resilience Scale (CD-RISC) validated by Laura with a=0.85). This will be measured by a scale as total scores and mean scores. High total and mean scores indicate better ability and readiness to take care giving responsibilities.
Quality of transition care among survivors and caregivers | within 1 month after discharge
  Quality of TC will be measured by the Care Transitions Measure (CTM) Tool developed by Eric Coleman. This will be measured by a scale as total scores and mean scores. High total and mean scores indicate better perceived quality of transition care.
Caregiver self-efficacy | 6 months after discharge
  Caregiver self-efficacy will be measured by the 10-items Family Caregiver Activation Tool (FCAT) developed by Coleman with a=0.6. This will be measured by a scale as total scores and mean scores. High total and mean scores indicate better ability to assist the stroke survivors to follow and adhere to healthy lifestyles and clinic appointment after stroke

SECONDARY OUTCOMES:
Depression and anxiety among survivors and caregivers | 6 months after discharge
  Depression and anxiety that will be measured by the locally validated 10-items Kessler Psychological Distress Scale with a=0.85. This will be measured by a scale as total scores and mean scores. High total and mean scores indicate poor mental health status after discharge.
Care satisfaction among survivors and caregivers | within 1 month after discharge
  Satisfaction of hospital care will be measured by a questionnaire developed specific for this study. It will be measured as total scores and mean scores. High total and mean scores indicate good satisfaction with transitional care.
Mortality among survivors | 6 months after discharge
  This will be counted as a death event after discharge.
readmission among survivors | 6 months after discharge
  This will be measured as number of times the patient is readmitted at the hospital after discharge. High frequency will indicate many readmissions.
length of hospital stay among survivors | Day 1 after discharge
  This will be measured as number of days spent in the hospital before discharge. This will be calculated as number of days spent at the hospital from admission to discharge. High number above 5 indicates long hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided
I will consider sharing it upon finishing enrollment of participants

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT07319312/Prot_SAP_ICF_000.pdf